CLINICAL TRIAL: NCT06499688
Title: A Randomized, Double-blind, Placebo- and Active-controlled Parallel-group Multi-center Phase III Study to Evaluate the Efficacy and Safety of Recombinant Botulinum Toxin Type A for Injection in the Treatment of Moderate to Severe Glabellar Lines
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of Recombinant Botulinum Toxin Type A for Injection in the Treatment of Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chongqing Claruvis Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YY001-001-Ⅲ-REFINE; CTR20233901 (Registry Identifier: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: YY001; Recombinant Botulinum Toxin Type A; Botulinum Toxin; Glabellar Lines
MeSH Terms: interventions — Injections; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Placebo- and active-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): Single injection with Rcombinant botulinum neurotoxin type A for injection(YY001) in glabellar lines
  Interventions: Biological: Rcombinant botulinum neurotoxin type A for injection (YY001)
- Active-Controlled Group (Active Comparator): Single injection with BOTOX® in glabellar lines
  Interventions: Biological: OnabotulinumtoxinA
- Placebo-Controlled Group (Placebo Comparator): Single injection with placebo in glabellar lines
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rcombinant botulinum neurotoxin type A for injection (YY001) — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.25 ml,0.05 ml per site.
  Arms: Treatment Group
Biological: OnabotulinumtoxinA — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.25 ml,0.05 ml per site.
  Arms: Active-Controlled Group
Biological: Placebo — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.25 ml,0.05 ml per site.
  Arms: Placebo-Controlled Group

SUMMARY:
This is a randomized, double-blind, placebo- and active-controlled parallel-group multi-center phase III study to evaluate the efficacy and safety of Rcombinant botulinum neurotoxin type A for injection (YY001)) in the treatment of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years (inclusive) at the time of signing the informed consent form.
2. At screening and baseline, moderate to severe glabellar lines (grade of 2 or 3 on the 4-point Scale) at maximal frown as assessed by both the Investigator and the participant on-site.
3. Agree to participate in the study and sign the informed consent form.
4. At the discretion of the investigator, the participants can comply with the protocol requirements.
5. Females and/or males of childbearing potential and their partners: those who should be using effective contraception and have no plans for childbearing, egg donation (females), or sperm donation (males) from the signing of the informed consent form to 3 months after the last administration. Female participants of childbearing potential must have had a negative blood pregnancy test (human chorionic gonadotropin) within 7 days prior to the administration of study drug or a urine pregnancy test examination must be negative 3 days prior to the administration of study drug.

Note:

1. Women of childbearing potential are those who have experienced menarche, have not undergone sterilization (hysterectomy or bilateral salpingo-oophorectomy or bilateral tubal ligation), and are not in a state of post-menopausal (defined as absence of menstrual bleeding for 12 months prior to screening, without any other medical reason).
2. Effective contraceptives include: vasectomy, abstinence, intrauterine devices, hormones [oral, patch, ring, injections, implants], barrier methods [diaphragm, cervical cap, sponge, condom.

Exclusion Criteria:

1. Known allergy to any component of the test product (includes investigational product and comparator product), or hypersensitivity.
2. Previous cosmetic manipulation of the area between the eyebrows, within 12 months prior to screening; implantation of autologous fat or any permanent material; history of upper face lifting or semi-permanent prosthetic fillers, etc.; or plan to undergo upper face cosmetic manipulation during the study period (note: except for study drug injections);
3. Use of any botulinum toxin within 6 months prior to baseline, or planned use of botulinum toxin during the study (note: except for use of investigational drugs at the study site).
4. Use of nonsteroidal anti-inflammatory drugs including aspirin or anticoagulants (e.g., heparin, coumarins, non-vitamin K antagonists, oral anticoagulants within 1 week prior to baseline.
5. Use of medications that affect neuromuscular transmission within 4 weeks prior to baseline, including but not limited to: muscarinic agents, aminoglycosides, anticholinergic agents, benzodiazepines.
6. At screening and baseline, skin abnormalities at the injection site
7. Inability to substantially lessen glabellar lines by physically spreading them apart, as determined by the investigator.
8. Ptosis, significant facial asymmetry, excessive skin laxity at screening or baseline, or a history of any of the above.
9. A history of facial nerve palsy.
10. History or presence of such diseases that interfere with neuromuscular function, including, but not limited to: myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis; diseases or a history of such diseases that can cause localized neuromuscular function, including, but not limited to: swallowing/breathing difficulties, diplopia, angle-closure glaucoma, significant drooping of the eyes and eyebrows, or flaccidity of the skin/excessive weakness or weakness of the corrugate and/or procerus;
11. Have other concomitant diseases, including but not limited to cardiovascular, respiratory, gastrointestinal, endocrine, and other systemic diseases, malignant tumors, and immunodeficiencies, which are assessed by the investigator to be unsuitable for participation in clinical research.
12. History of drug or alcohol abuse.
13. History or presence of epilepsy.
14. Female who is pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The 4th week after treatment, the composite response rate on both the investigator's assessment and the participant's self-assessment concurrently of GL severity at maximal frown. | The 4th week after treatment
  The composite response rate: The proportion of participants achieving a score of 0 or 1 and a two-grade improvement from the baseline, on both the investigator's assessment and the participant's self- assessment concurrently of GL severity at maximal frown.
  Glabellar lines at maximal frown is based on the 4 grade Facial Wrinkle Scale: 0 (none), 1 (mild), 2 (moderate) and 3 (severe).
At the 1st week, 8th week, and 12th week after treatment, the composite response rate on both the investigator's assessment and the participant's self- assessment concurrently of GL severity at maximal frown. | At the 1st week, 8th week, and 12th week after treatment

SECONDARY OUTCOMES:
The response rate on the investigator's assessment and the participant's self- assessment individually of GL severity at maximal frown and the Independent Review Committee's assessment of GL severity photos at maximal frown taken on-site. | At the 1st week, 4th week, 8th week, and 12th week after treatment
  The response rate: The proportion of participants achieving a score of 0 or 1 and a two-grade improvement of GL severity from the baseline at maximal frown.
The proportion of participants who achieve a score of 0 or 1 on the investigator's assessment and the participant's self-assessment individually of GL severity at maximal frown and the Independent Review Committee's assessment. | At the 1st week, 4th week, 8th week, and 12th week after treatment
  The proportion of participants who achieve a score of 0 or 1 on the investigator's assessment and the participant's self-assessment individually of GL severity at maximal frown and the Independent Review Committee's assessment of GL severity photos at maximal frown taken on-site.
the severity of GL at rest on the investigator's assessment and the participant's self- assessment individually of GL severity at maximal frown and the Independent Review Committee's assessment of GL severity photos at maximal frown taken on-site. | At the 1st week, 4th week, 8th week, and 12th week after treatment
  The severity of glabellar lines at rest will be assessed according to the 4 grade scale: 0 (none), 1 (mild), 2 (moderate) and 3 (severe).
The duration of GL treatment effect when the maximal frown severity score returned to baseline score. | Within 12 weeks
At the 1st week, 4th week, 8th week, and 12th week after treatment, the improvement rate of glabellar lines severity at maximal frown on the participant's self-assessment. | At the 1st week, 4th week, 8th week, and 12th week after treatment
  Participant self-assessment of 9 subscales: +4 (complete improvement), +3 (significant improvement), +2 (moderate improvement), +1 (slight improvement), 0 (no change), -1 (minor aggravation), -2 (medium aggravation), -3 (significant aggravation), and-4 (very significant aggravation).
  Improvement rate is defined as the proportion of participants with + 2 (moderate improvement) or above.
At the 1st week, 4th week, 8th week, and 12th week after treatment, the participant's satisfaction. | At the 1st week, 4th week, 8th week, and 12th week after treatment
  Satisfaction will be assessed on the 7-grade scale: 1 (very dissatisfied), 2 (dissatisfied), 3 (somewhat dissatisfied), 4 (reluctantly), 5 (relatively satisfied), 6 (satisfied) and 7 (very satisfied).
  Calculate the proportion of participants with 6 or above.
Incidence of adverse events and serious adverse events within 12 weeks of treatment. | Within 12 weeks of treatment
Incidence of injection site reactions within 12 weeks of treatment. | Within 12 weeks of treatment
Incidence of anti-drug antibodies and neutralizing antibodies within 12 weeks of treatment. | Within 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wu, Principal Investigator — Peking University First Hospital
Locations (16):
- China (16):
  - Guangdong Second People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xian, Shanxi
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hangzhou First People's Hospital, Westlake University, School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking Union Medical College Hospital , Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Plastic Surgery Hospital, Chinese Academy of Medical Science, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No